CLINICAL TRIAL: NCT04716452
Title: Phase I Study of C6 Ceramide NanoLiposome (CNL) in Patients With Relapsed/Refractory Acute Myeloid Leukemia (RR-AML)
Brief Title: Study of C6 Ceramide NanoLiposome (CNL) in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Acronym: KNAN2001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Keystone Nano, Inc (Industry)
Collaborators: University of Virginia (Other); Milton S. Hershey Medical Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNAN2001; 5R44CA275609-02 (NIH)
Record Dates: First submitted 2020-11-30; First posted 2021-01-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia, Refractory; Refractory/Relapse Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Relapsed; Refractory; Ceramide; AML; NanoLiposome; Relapsed/Refratory Acute Myleoid Leukemia; NanoLiposomes; Safety
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Administration of Ceramide NanoLiposome (Experimental): Ceramide NanoLiposome will be administered by Intravenous Dosing twice per week in accordance with the protocol relative to dose escalation. There is no placebo group or arm of the study.
  Interventions: Drug: Ceramide NanoLiposome (Ceraxa)

INTERVENTIONS:
Drug: Ceramide NanoLiposome (Ceraxa) — Ceramide NanoLiposome will be given by IV twice a week. The dose, which is based on body size, will be increased for the next group of patients if the first group of patients tolerates that dose and it will decrease for the next group if they do not tolerate the dose.
  Other Names: Ceramide NanoLiposome

SUMMARY:
The study objective is to evaluate patient safety for patients with refractory and relapsed AML being treated with Ceramide NanoLiposome (CNL) .

DETAILED DESCRIPTION:
The research team has shown that C6 ceramide nanoliposome (CNL) has anti-cancer activity in laboratory models of AML and that when it is combined with other cancer-fighting drugs, it works better.

The primary goal of this study is to evaluate the safety of CNL given without other cancer treatments in patients with AML where either their initial treatment didn't work or it stopped working and the AML came back (refractory or relapsed AML, aka RR-AML). This study seeks to determine the right dose to start with in later studies when CNL is combined with other drugs in potential future studies.

CNL is given by intravenous (IV) infusion and will be given twice a week in this study. Participants will receive study treatment as long as it is considered safe for them to continue, though their disease status will be checked regularly to make sure that their disease has not gotten worse. Blood samples will be collected at many time-points to see how their bodies are responding to the drug and how long it stays in the blood.

The first patients in the study will start at one dose of the drug and, if that is shown to be safe, the next group will be treated at a slightly higher dose. Participants will be given CNL by intravenous (IV) infusion twice a week over about 2 hours and then they will be monitored for about 2 hours to make sure they don't have any bad side effects, but initially patients will be required to stay at the site for about 6 hours after the start of the infusion in order to get blood draws to see how long the drug stays active in their system.

Participants will have a bone marrow biopsy before their second "cycle" of drug (after about 1 month) and then again before their third cycle of drug in order to see how their disease is responding. After that, bone marrow biopsies will be about every other cycle based on what the study doctor recommends. If the doctor doesn't think that CNL is helping their disease, or if their doctor decides that it is not safe for them to continue, they will be taken off study treatment. Participants will be followed for safety and disease status for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent is obtained prior to conducting any study-specific screening procedures.
2. Willing and able to understand the nature of this study and to comply with the study and follow-up procedures.
3. Age and Disease: ≥ 18 years of age with refractory or relapsed AML

   Refractory AML: Patients who fail to achieve a complete remission (CR) after one line of AML directed therapy

   Relapsed AML: Patients who achieved a complete remission (CR) with one or more prior lines of AML directed therapy but then developed a relapse of AML.

   Note: Patients are eligible even if they have not received intensive induction chemotherapy but have been treated with other AML directed therapy like hypomethylating agents (azacitidine, decitabine).
4. Eastern Cooperative Oncology Group (ECOG) performance status must be ≤2
5. Peripheral white blood cell (WBC) count <30,000/µL. For cyto-reduction, hydroxyurea is allowed during screening and through Cycle 2, Day 3 to reduce WBC count to < 30,000 µL.
6. Adequate organ function as evidenced by the following laboratory findings:

   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN) or < 3 x ULN for patients with Gilbert-Meulengracht Syndrome
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN
   * Creatinine clearance > 60 mL/min
7. QT-interval corrected according to Fridericia's formula (QTcF) < 450 ms on one electrocardiogram (ECG) at screening

Exclusion Criteria:

Patients meeting any of the following criteria are ineligible for study entry:

1. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmias not well controlled with medication, myocardial infarction within the previous 6 months before registration, or psychiatric illness/social situations that would limit compliance with study requirements.
2. Patients may not be receiving any other concurrent investigational agents, or have received any investigational agent within one week of registration.
3. Since the teratogenic potential of this combination is currently unknown, females who are pregnant or lactating are excluded.
4. History of any other malignancies within the preceding 12 months before registration with the exception of in-situ cancer, non-muscle invasive bladder cancer, prostate, basal or squamous cell skin cancer
5. Life-threatening illnesses other than AML, uncontrolled medical conditions or organ system dysfunction that, in the Investigator's opinion, could compromise the patient's safety or put the study outcomes at risk
6. Evidence of isolated extramedullary disease
7. Acute Promyelocytic Leukemia or AML with active central nervous system (CNS) involvement
8. Untreated severe (in the opinion of the treating investigator) infection
9. Active and uncontrolled infection with HIV (viral load is detectable by PCR)
10. Active infection with Hepatitis B virus (HbSAg positive or PCR with detectable viral load) or Hepatitis C virus (viral load detectable by PCR).
11. Past Hematopoietic stem cell transplant (HSCT) with active graft vs host disease, immunosuppression other than low dose prednisone (5 mg), or calcineurin inhibitors within the 4 weeks before registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicities as defined in Protocol Section 13.5 | At the end of the the first cycle of administration (each cycle is 28 days)
  Dose Limiting Toxicities within the first cycle of CNL monotherapy. See section 13.5 of Protocol for the complete list of Dose Limiting Toxicities
Number of Patients with Adverse Events | Through study completion, an average of 24 weeks
  Number of Patients with Adverse Events
Severity of Adverse Events | Through study completion, an average of 24 weeks
  Severity of Adverse Event As Described in Protocol
Duration of Adverse Events | Length of Adverse Events as measured in days, measured through study completion, an average of 24 weeks
  Duration of Adverse Events, As Described in Protocol, measured in days
Duration of therapy | Through study completion, an average of 24 weeks
  Duration of therapy provided as measured in days
Dose Levels achieved during study | Through study completion, an average of 24 weeks
  Dose levels administered in milligrams per m2
Concentration Max (C Max) | Through cycle one, 28 days (each cycle is 28 days)
  Maximum Serum Concentration measured, in nanograms/milliliter
Time to Maximum Study Drug (T Max) | Through cycle one, 28 days (each cycle is 28 days)
  Time to maximum concentration measured, in minutes
Half Life of Study Drug | Through cycle one, 28 days (each cycle is 28 days)
  Time for drug to be reduced to half of the starting concentration (in minutes)
Study Drug Clearance | Through cycle one, 28 days (each cycle is 28 days)
  The Amount of Study Drug Cleared per unit time (Nanograms/Minute)
Ratio of C16/C24 Ceramides | After one cycle of therapy (Day 28)
  Ratio of Ceramide 16 to Ceramide 24 (ng of C16/ng of C18) from bone marrow biopsy
Clinical Response - Complete Response | After Cycle Two (56 days)
  Complete Response
Clinical Response - Complete Response with Incomplete Hematologic Recovery (CRi) | After Cycle Two (56 days)
  Complete Response with Incomplete Hematological Recovery as defined by blasts in bone marrow
Clinical Response - Partial Remission | After Cycle Two (56 days)
  Partial Remission (as defined by blasts in bone marrow)

SECONDARY OUTCOMES:
Number of Patients with Grade 3 or 4 Adverse Events | Through study completion, an average of 24 weeks
  Grade 3 and 4 adverse events as defined by CTCAE v5.0
Overall Response | Through study completion, an average of 24 weeks, and up to 24 weeks afterwards (total of 48 weeks)
  Overall response of CNL monotherapy in patients with RR-AML: Complete remission (CR) + Complete remission with incomplete count recovery (CRi) + partial response (PR). CR, CRi and PR as defined as European LeukemiaNet 2017 (ELN 2017) response criteria
Event Free Survival | From registration to 24 weeks after completion of experimental drug treatment
  Event-free survival (EFS): the time from registration until documented refractory disease, relapse after achieving CR/CRi, or death from any cause, whichever is observed first
Overall Survival | From registration to 24 weeks following drug administration
  Overall survival (OS)
Quality of Life according to EORTC Quality of Life Questionnaire (QLQ) C30 | Prior to starting study treatment, on day 1 of each cycle (each cycle is 28 days), and at end of treatment (which is expected to be 2 to 3 months (cycles) for most patients
  Quality of life according to EORTC Quality of Life Questionnaire C30

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Vlock, MD, Study Director — Keystone Nano, Inc; Christopher Prior, Ph.D., Study Chair — Keystone Nano
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Likely to be shared with PO1 Researchers at UVA and Penn State. In addition to yearly FDA reports, anticipate potential manuscripts as well but not yet decided with all participants.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Dec 1, 2026
Access Criteria: 6 months after Trial

REFERENCES:
- [Background] Barth BM, Wang W, Toran PT, Fox TE, Annageldiyev C, Ondrasik RM, Keasey NR, Brown TJ, Devine VG, Sullivan EC, Cote AL, Papakotsi V, Tan SF, Shanmugavelandy SS, Deering TG, Needle DB, Stern ST, Zhu J, Liao J, Viny AD, Feith DJ, Levine RL, Wang HG, Loughran TP Jr, Sharma A, Kester M, Claxton DF. Sphingolipid metabolism determines the therapeutic efficacy of nanoliposomal ceramide in acute myeloid leukemia. Blood Adv. 2019 Sep 10;3(17):2598-2603. doi: 10.1182/bloodadvances.2018021295. PMID 31488436
- [Background] Morad SAF, MacDougall MR, Abdelmageed N, Kao LP, Feith DJ, Tan SF, Kester M, Loughran TP Jr, Wang HG, Cabot MC. Pivotal role of mitophagy in response of acute myelogenous leukemia to a ceramide-tamoxifen-containing drug regimen. Exp Cell Res. 2019 Aug 15;381(2):256-264. doi: 10.1016/j.yexcr.2019.05.021. Epub 2019 May 18. PMID 31112736
- [Background] Kester M, Bassler J, Fox TE, Carter CJ, Davidson JA, Parette MR. Preclinical development of a C6-ceramide NanoLiposome, a novel sphingolipid therapeutic. Biol Chem. 2015 Jun;396(6-7):737-47. doi: 10.1515/hsz-2015-0129. PMID 25838296